CLINICAL TRIAL: NCT07133438
Title: Mecobalamin Combined With Anti-VEGF Intravitreal Injection for Treatment Retinal Vein Occlusion: a Double-blind Randomized Controlled Trial
Brief Title: Mecobalamin Combined With Anti-VEGF Intravitreal Injection for Retinal Vein Occlusion Treatment
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yan-Lai Zhang, associate chief physician, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: No. 2025-387-01
Record Dates: First submitted 2025-06-29; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Retinal Vein Occlusion (RVO)
Keywords: Retinal Vein Occlusion (RVO); Macular edema; Anti-VEGF
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — mecobalamin

STUDY DESIGN:
Intervention Model Description: a double-blind randomized controlled trial
Who Masked: Participant, Investigator
Masking Description: All study participants will be blinded to their intervention assignment. The drug and placebo were identical in packaging, appearance, and smell. Mecobalamin and placebo were assigned by an independent pharmacy according to random codes. Evaluators were blinded to group allocation. All study medications (active and placebo) will be identically labeled to ensure adequate blinding of study physicians and patients. Patients, principal investigators, assessor physicians, imaging technicians, central reading center graders, study coordinators, and BCVA examiners will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): Patients in the experimental group will receive conventional anti-VEGF therapy (intravitreal injections of conbercept 0.5 mg initially once a month for 3 months, followed by on-demand therapy which based on recurrence criteria) along with oral mecobalamin capsules 0.5 mg three times daily for 6 months.
  Interventions: Drug: Anti-VEGF drug; Drug: Mecobalamin 5 MG
- control group (Placebo Comparator): Patients in the control group will receive the same anti-VEGF treatment as the experimental group and will take a placebo capsule with a similar appearance and odor to the mecobalamin capsules three times daily for 6 months
  Interventions: Drug: Anti-VEGF drug; Drug: Placebo

INTERVENTIONS:
Drug: Anti-VEGF drug — conventional anti-VEGF therapy (intravitreal injections of conbercept 0.5 mg initially once a month for 3 months, followed by on-demand therapy which based on recurrence criteria)
Drug: Mecobalamin 5 MG — oral mecobalamin capsules 0.5 mg three times daily for 6 months
  Arms: experimental group
Drug: Placebo — placebo capsule with a similar appearance and odor to the mecobalamin capsules three times daily for 6 months
  Arms: control group

SUMMARY:
Retinal vein occlusion (RVO), a common retinal vascular disease, is frequently treated with anti-vascular endothelial growth factor (anti-VEGF) agents as first-line therapy. However, anti-VEGF monotherapy lacks neuroprotective effects, primarily targets vascular leakage and neovascularization, and requires frequent long-term injections that impose substantial economic burdens. Combined therapeutic strategies addressing both vascular pathology and neural damage are therefore being explored.

This article describes the protocol for a randomized, outcome-blinded, placebo-controlled clinical trial evaluating mecobalamin (a widely used neuroprotective drug) in combination with anti-VEGF for the treatment of macular edema (ME). A total of 120 eligible RVO patients will be enrolled from the First Affiliated Hospital of Chongqing Medical University. Participants will be randomly assigned (1:1) to an experimental group and a control group. The experimental group will receive conventional anti-VEGF therapy plus oral mecobalamin capsules for 6 months, while the control group will receive the same anti-VEGF treatment plus a placebo for 6 months. All patients will undergo one year of follow-up after initial treatment, with visits at 1, 3, 6, 9, and 12 months.

The primary outcome is the change in central foveal thickness (CFT) from baseline to one year post-initial treatment. Secondary outcomes include:

* Change in best-corrected visual acuity (BCVA) from baseline over time,
* Capillary density,
* Cone photoreceptor distribution characteristics,
* Mean light sensitivity and fixation stability,
* Serum vitamin B12 levels,
* Number of anti-VEGF treatments,
* Injection frequency (times per year),
* Treatment interval,
* Incidence and severity of adverse events (AEs) and serious adverse events (SAEs).

This trial evaluates a novel "neuroprotection + vascular intervention" strategy combining mecobalamin with anti-VEGF therapy. The trial aims to provide high-level evidence for synergistic RVO treatment, with the potential to reduce recurrence rates and improve long-term visual function prognosis.

DETAILED DESCRIPTION:
Retinal vein occlusion (RVO) is the second leading cause of vision loss resulting from retinal vascular disease, with a prevalence of approximately 0.6%-1.6%. Macular edema (ME) secondary to RVO is a common cause of vision loss. RVO induces hypoxia and ischemia, leading to neuronal loss and increased vascular permeability. Therefore, anti-vascular endothelial growth factor (anti-VEGF) injections are widely used as first-line treatment for RVO-ME, achieving remarkable therapeutic effects. Pivotal trials (BRAVO and CRUISE) demonstrated that anti-VEGF therapy significantly improves best-corrected visual acuity (BCVA) and reduces retinal swelling, enhancing BCVA by 12-15 ETDRS letters and decreasing central foveal thickness (CFT) by about 200 μm.

However, therapies targeting VEGF alone may not sufficiently manage this condition. Although anti-VEGF agents improve edema and short-term visual acuity, long-term efficacy is limited by frequent injections and inadequate nerve repair. Additionally, anti-VEGF fails to reverse neurodegenerative changes such as photoreceptor apoptosis and Müller cell activation. Consequently, combined strategies synchronizing vascular leakage repair and neuroprotection have become an international research priority.

As a typical neurotrophic drug, mecobalamin repairs nerve tissue and accelerates axonal regeneration and myelination. Mecobalamin, a vitamin B12 derivative, is more readily absorbed by nerve cells than vitamin B12 itself. As a methyl donor, it facilitates homocysteine-to-methionine conversion, supporting nucleic acid, protein, and phospholipid synthesis critical for myelin formation. This process is essential for nerve myelin formation and repair. Mecobalamin accelerates lipid, protein, and nucleic acid metabolism in neurons, enhancing nerve function recovery and alleviating neurological symptoms. Previous studies found that oral vitamin B1 and mecobalamin improve corneal nerve fiber density. The neuroprotective drug was shown to attenuate oxidative stress in animal models, but clinical translation evidence remains insufficient.

Notably, VEGF exhibits dual roles as both a permeability factor and neuroprotectant. Excessive VEGF inhibition may exacerbate retinal ganglion cell apoptosis. Although mecobalamin promotes neural repair, its spatiotemporal synergy with anti-VEGF in neurovascular unit (NVU) recovery remains uncharacterized. This prospective, double-blind, randomized controlled trial evaluates the synergistic effects of mecobalamin combined with anti-VEGF therapy on NVU repair in RVO-ME, utilizing dual-targeted "vascular intervention + neuroprotection" to overcome current limitations.

Current ME efficacy assessment relies primarily on optical coherence tomography (OCT)-derived CFT, with few tertiary centers employing OCT angiography (OCTA), multifocal electroretinography (mfERG), or adaptive optics (AO). Existing metrics inadequately characterize NVU function or anti-VEGF effects on non-vascular components (glia, photoreceptors). The absence of standardized NVU repair quantification impedes cross-study comparisons. To address this, the investigators propose a multimodal "OCT structural tomography + OCTA flow stratification + AO cellular morphology + microperimetry functional mapping + mfERG functional localization" assessment to establish a new therapeutic standard.

Primary objectives:

1. Evaluate mecobalamin combined with anti-VEGF therapy on CFT and BCVA improvement in RVO-ME patients
2. Validate mecobalamin's synergistic contribution to NVU repair using multimodal imaging

This prospective, double-blind, randomized controlled intervention study will enroll RVO patients at the First Affiliated Hospital of Chongqing Medical University from 1 August 2025 to 31 July 2027. The study aims to evaluate mecobalamin combined with conbercept on retinal NVU repair in RVO-ME patients. The Institutional Review Board approved the protocol (No. 2025-387-01) on 26 May 2025. The study adheres to the Declaration of Helsinki and Ethical Guidelines for Medical and Biological Research Involving Human Subjects. All participants will provide written informed consent; an opt-out approach will be implemented where applicable.

Primary outcomes will be assessed at 12 months post-initial treatment. Eligible patients will be identified during initial ophthalmology visits. Recruitment will be performed by ophthalmologists. After eligibility confirmation and informed consent, standard treatment commences immediately. Reasons for non-participation will be documented. Enrolled eyes will receive alphanumeric ID codes and be randomly assigned to treatment groups two days before intervention using block randomization (Statistical Package R, v3.6).

Treatment groups (1:1 randomization):

Experimental: Intravitreal conbercept (0.5 mg monthly × 3 months, then pro re nata) + oral mecobalamin (0.5 mg TID × 6 months) Control: Identical anti-VEGF regimen + placebo capsules (TID × 6 months)

Recurrence criteria:

* CFT increase ≥50 μm from minimum recorded value
* BCVA decrease ≥5 ETDRS letters
* New/increased intraretinal/subretinal fluid

Assessments occur at baseline, initial treatment day, and 1, 3, 6, 9, and 12 months post-treatment. Follow-up requirements are detailed in supplementary materials. Study exit occurs at 1-year completion or if:

1. Three consecutive missed visits
2. Poor compliance/withdrawal request
3. New systemic disease affecting outcomes

Protocol violators or cases with essential missing data will be excluded from per-protocol analysis. Clinical trial staff will collect data under investigator supervision. Researchers will ensure data accuracy, completeness, and timeliness. The schedule for enrollment, interventions, and assessments is outlined in supplementary materials. Clinical/ophthalmic data will be entered into an electronic data capture system. All data will remain confidential per regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of RVO meeting the international diagnostic criteria 4,12, age 18-80 years, gender not limited Treatment-naive RVO-ME (no prior anti-VEGF, glucocorticoid, or laser therapy) The CFT is confirmed to be ≥300μm by OCT The baseline BCVA (ETDRS letter count) was 20/400 to 20/40 (34-78 letters) Signed informed consent and ability to comply with follow-up.

Exclusion Criteria:

Combined with other eye diseases that cause ME (such as diabetic retinopathy, uveitis) Media opacities affecting imaging (such as severe cataract, vitreous hemorrhage) Prior anti-VEGF, steroid, or macular laser therapy Systemic use of glucocorticoids or immunosuppressants within 3 months Uncontrolled systemic disease (hypertension, diabetes, hepatic/renal dysfunction); pregnant or lactating women Allergy to mecobalamin or conbercept Unable to cooperate with examinations or follow-up, or participate in other clinical trials within one year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Anatomical indicators-central foveal thickness | From enrollment to the end of treatment at 1 year
  the changes in central foveal thickness from baseline to 1 year post initial treatment.The primary outcome is the change in central foveal thickness (CFT), measured via spectral-domain optical coherence tomography (SD-OCT), from baseline to 12 months post-initial treatment. CFT will be defined as the mean retinal thickness within the central 1-mm diameter subfield of the ETDRS grid (Early Treatment Diabetic Retinopathy Study), automatically segmented and calculated using device software (e.g., Heidelberg Spectralis® or equivalent). All OCT scans will be performed by certified technicians following standardized protocols, including quality control for signal strength (>7/10), proper centering, and absence of artifacts. Measurements will be verified by masked graders at a central reading center.

SECONDARY OUTCOMES:
Change in best-corrected visual acuity (BCVA) | From enrollment to the end of treatment at 1 year
  Change in best-corrected visual acuity (BCVA) from baseline over time (months 1,3,6,9,12), assessed using ETDRS charts at 4 meters under standardized luminance (85-120 cd/m²). BCVA will be quantified as letters read (0-100 scale) following manifest refraction, with scoring adherence to ETDRS standards. All measurements will be performed by masked examiners with central reading center quality control.
capillary density | From enrollment to the end of treatment at 1 year
  Changes in capillary density, assessed as vessel density (%) in the superficial and deep retinal capillary plexuses using optical coherence tomography angiography (OCTA). Scans will be acquired with a standardized 3×3 mm or 6×6 mm pattern centered on the fovea, processed with projection artifact removal, and quantified within ETDRS grid subfields. All analyses will undergo quality control and centralized grading.
cone photoreceptor density | From enrollment to the end of treatment at 1 year
  Changes in cone photoreceptor density (cones/mm²) assessed using adaptive optics ophthalmoscopy centered at the fovea. Images will be processed with semi-automated cone identification algorithms and compared against normative databases. All analyses require dual masked grading with quality control (Strehl ratio ≥0.2, SNR >25 dB).
the mean light sensitivity | From enrollment to the end of treatment at 1 year
  Changes in mean light sensitivity (dB) assessed using microperimetry (68-point central 10° grid, 4-2 staircase strategy) under standardized conditions. Testing requires pupil dilation ≥6 mm, with validity criteria including <15% false-positive rate and <20% fixation losses. All analyses will undergo central reading center verification.
Serum vitamin B12 levels | From enrollment to the end of treatment at 1 year
  Changes in serum vitamin B12 levels, measured via chemiluminescent microparticle immunoassay (CMIA) on fasting morning samples. Testing will follow standardized pre-analytical protocols with ARCHITECT® or Cobas® platforms. Results will be interpreted against WHO reference ranges (deficiency: <200 pg/mL) with quality control criteria including CV ≤5% and linearity R²≥0.99.
the number of treatments | From enrollment to the end of treatment at 1 year
  Total anti-VEGF treatments: Cumulative intravitreal injections over 12 months
incidence of adverse events (AEs) | From enrollment to the end of treatment at 1 year
  AEs incidence:Proportion of participants with ≥1 event, categorized by system organ class (MedDRA) and severity (CTCAE v6.0/OTS)
incidence of serious adverse events (SAEs) | From enrollment to the end of treatment at 1 year
  SAEs incidence:Proportion of participants with ≥1 event, categorized by system organ class (MedDRA) and severity (CTCAE v6.0/OTS)

CONTACTS AND LOCATIONS:
Locations (1):
- No. 1, Friendship Road, Yuanjiagang, Yuzhong District, Chongqing City, Chongqing, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol